CLINICAL TRIAL: NCT00179738
Title: A Multicenter, Single-Arm, Open-Label, Study To Evaluate The Safety And Efficacy Of Single-Agent Lenalidomide (Revlimid®) In Subjects With Androgen Independent Prostate Cancer
Brief Title: A Multicenter, Single-Arm, Open-Label, Study to Evaluate the Safety and Efficacy of Single-Agent Lenalidomide (Revlimid, CC-5013) in Subjects With Androgen Independent Prostate Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: Prologue Research International (Industry)
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-PC-001
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2005-09

CONDITIONS: Prostate Cancer
Keywords: Androgen Independent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lenalidomide

INTERVENTIONS:
Drug: CC5013

SUMMARY:
Subjects who qualify will receive single agent oral lenalidomide daily on days 1-21 every 28 day cycle. Subjects will continue on study until documented disease progression

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age > or = to 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Must have a histologic diagnosis of adenocarcinoma of the prostate.
5. Must be surgically or medically castrated. If the method is medical castration, the subject must have a serum testosterone level of <50 ng/dl. The subject should maintain treatment with LH RH antagonists or agonists.
6. Must have prostate cancer unresponsive or refractory to androgen blockade as demonstrated by rising PSA.

   -Rising PSA is defined as at least 2 consecutive rises in PSA to be documented over the reference value (measure 1). The first rising PSA (measure 2) must be taken at least 7 days after the reference value.

   A third confirmatory PSA is required, and it must be obtained at least seven days after the second measure. If this is not greater than measure 2, a fourth PSA is required and this must be greater than measure 2.

   -Absolute value of PSA > or = to 5 ng/ml on the last confirmatory assessment.
7. Prior treatment with antiandrogens such as flutamide, or other hormonal agents such as estrogens, corticosteroids, or ketoconazole must have been stopped for at least 28 days prior to treatment.

   In the case of nilandron and bicalutamide, treatment with these agents must have stopped at least 42 days prior to treatment. Following completion of the antiandrogen withdrawal period, either:
   * One post withdrawal PSA value must be higher than the last pre-withdrawal PSA value, or
   * If the subject's PSA value decreased following the antiandrogen withdrawal period then two increases in PSA values must be documented after the post-withdrawal nadir.
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 (Appendix II: ECOG Performance Status Scale).

Exclusion Criteria:

1. Metastatic prostate cancer
2. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) <1,500 cells/mm3 (1.5 x 109/L)
   2. Platelet count <100,000 cells/mm3 (100 x 109/L)
   3. Serum creatinine >2.5 mg/dL (221 mmol/L)
   4. Serum SGOT/AST or SGPT/ALT >3.0 x upper limit of normal (ULN)
   5. Serum total bilirubin >2.0 mg/dL (34 mmol/L)
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study or confounds the ability to interpret data from the study.
4. Prior history of malignancies other than AIPC (except for basal cell or squamous cell carcinoma of the skin) unless the subject has been free of the disease for > or = to 1 year.
5. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
6. Prior > or = to grade 3 allergic reaction/hypersensitivity to thalidomide.
7. Prior > or = to grade 3 rash or any desquamating (blistering) rash while taking thalidomide.
8. Prior use of lenalidomide.
9. Prior use of chemotherapy for androgen independent prostate cancer.
10. Use of any standard/experimental anti-cancer drug therapy within 28 days of the initiation of study drug therapy except LHRH agonists/antagonists.
11. Known active Hepatitis C.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-04; Study Completion 2007-04

PRIMARY OUTCOMES:
To determine the activity of lenalidomide monotherapy in subjects with androgen independent prostate cancer (AIPC).

SECONDARY OUTCOMES:
To evaluate the safety of lenalidomide monotherapy as treatment for subjects with AIPC.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Alta Bates Cancer Center, Berkeley, California
  - Moffit Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Seattle Cancer Care Alliance, Seattle, Washington